CLINICAL TRIAL: NCT02168452
Title: Clinical Application of Dual Sentinel Lymph Node Staining Method in Breast Cancer Patients Who Receive Neoadjuvant Chemotherapy; Observational Pilot Study
Brief Title: Clinical Application of Dual Sentinel Lymph Node Staining Method in Breast Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Seeyoun Lee, Medical Doctor, National Cancer Center, Korea
Other Study IDs: NCC-1410201-1
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant chemotherapy; Indocyanine green (ICG); Radioisotope (RI); Near infrared fluorescence camera
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: sentinel lymph node biopsy(SLNB) — * incision will be made over the skin site that had fluorescence lymphatic flow which visualized using fluorescence imaging camera and gamma probe.
  * double check after removal of the sentinel lymph node
  * sending frozen biopsy

SUMMARY:
This study aimed to evaluate the feasibility of dual sentinel node staining method using mixture of indocyanine green(ICG) and radioisotope (RI) in breast cancer patients who receive neoadjuvant chemotherapy.

Over the past few years, several studies have found using methylene blue, isosulfan blue, indocyanine green or radioisotope alone by detection method had several disadvantages.

In this study we expects using mixture of indocyanine green (ICG) with radioisotope (RI) has potential to improve sentinel lymph node (SLN) mapping in breast cancer patients who receive neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
* 5 patients who receive neoadjuvant chemotherapy with cN1-cN2 or cT2 on TNM staging
* sentinel lymph node biopsy(SLNB) by sentinel lymph node staining method using mixture of indocyanine green (ICG) with radioisotope (RI).
* indocyanine green (ICG) penetrates human tissue to depths of several millimeters to 2cm, and the fluorescence can be detected percutaneously in real time.
* using RI only has several disadvantages such as invisibility,interference. RI only detect sound or confirm numerical value through gamma probe.
* ICG can be visualized with a fluorescence imaging system
* confirm Identification rate of sentinal lymph node biopsy, and duration of sentinel lymph node biopsy

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients who receive neoadjuvant chemotherapy
* cN1-cN2 or cT2 on tumor lymphnode metastasis classification(TNM)
* ECOG Performance status 0 or 1
* consented patients with more than 20 years, less than 70 years

Exclusion Criteria:

* history of breast cancer
* early stage breast cancer
* history of excisional or incisional biopsy or axillary dissection
* inflammatory breast carcinoma
* cN3 on tumor lymphnode metastasis classification(TNM)
* history of hormone therapy or targeted therapy
* stage 4 breast cancer
* pregnancy

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who receive neoadjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Identification rate of sentinal lymph node biopsy | during operation
  It was defined as the ability to identify a sentinel lymph node successfully.

SECONDARY OUTCOMES:
duration of sentinel lymph node biopsy | during operation
  It was defined as the time from the skin incision to complet removal of the first sentinel lymph node.

OTHER OUTCOMES:
Physical assess | follwing up a week to 3month
  * assess pigmented skin lesion
  * assess for other complication

CONTACTS AND LOCATIONS:
Overall Officials: Seeyoun Lee, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea